CLINICAL TRIAL: NCT04069416
Title: Salvage Living Donor Liver Transplantation for HCC Beyond All Criteria Yield Equivalent Results to Milan Criteria in High Prevalence Young HCC Patients Country.
Brief Title: Salvage Living Donor Liver Transplantation for HCC Beyond All Criteria Yield Equivalent Results to Milan Criteria
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manar Salah, Principal investigator, Ain Shams University
Other Study IDs: 68954200
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hcc
Keywords: liver transplant; HCC; Extended milan; Living donor liver transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 175 patients who fall within the Milan criteria.
  Interventions: Procedure: living donor liver transplantation
- Group II: 36 patients who fall within up-to-7 criteria
  Interventions: Procedure: living donor liver transplantation
- Group III: 30 patients beyond up-to-7 criteria and will be termed beyond all criteria (BAC).
  Interventions: Procedure: living donor liver transplantation

INTERVENTIONS:
Procedure: living donor liver transplantation — liver graft from a living donor

SUMMARY:
The present study aims to evaluate the impact of expanding criteria beyond Milan on tumor recurrence and patient survival that will help identify the best selection criteria for HCC transplanted patients.

DETAILED DESCRIPTION:
Introduction:

HEPATOCELLULAR CARCINOMA (HCC) is the second leading cause of cancer mortality worldwide. Living donor liver transplantation (LDLT) for HCC patients has emerged as a rewarding therapy for a cure and a successful alternative where a Deceased donor liver transplantation (DDLT) program is lacking. Therefore, trials for careful expansion to Milan criteria have been adopted.

Aim of the study:

To evaluate the impact of expanding criteria beyond Milan on tumor recurrence and patient survival that will help identify the best selection criteria for HCC transplanted patients

ELIGIBILITY:
Inclusion Criteria:

* All patient transplanted for HCC eligible for transplant (no vascular invasion-no extra hepatic metastasis)
* age>18y

Exclusion Criteria:

* other etiology for liver transplant rather than HCC
* patient not fit for surgery
* age >70y

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were divided according to the pre-transplant radiological findings of HCC nodules number and sizes into 3 groups:
  Group I: comprised 175 patients who fall within the Milan criteria. Group II: included 36 patients who fall within up-to-7 criteria (the sum of the number of the tumors and diameter of the largest tumor not exceeding 7cm) Group III: included 30 patients beyond up-to-7 criteria and will be termed beyond all criteria (BAC).
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
HCC recurrence | 3 years
  Recurrence of Hepatocellular carcinoma either intra-hepatic, extra-hepatic or both

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol